CLINICAL TRIAL: NCT00071617
Title: Youth Support Team Intervention for Suicidal Adolescents
Brief Title: Youth-Nominated Support Team Intervention for Suicidal Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Cheryl A. King, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH063881 (NIH); R01MH063881 (NIH); DSIR 84-CTS
Record Dates: First submitted 2003-10-29; First posted 2003-10-30 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Suicide, Attempted
Keywords: Suicide; Adolescence
MeSH Terms: conditions — Suicide, Attempted; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Youth-Nominated Support Team (Experimental): Adolescents nominate up to 4 caring adults from family, school, community settings. These adults participate in psychoeducation sessions regarding adolescent's treatment plan and support needs. They maintain regular, supportive contact with the adolescent for 3 months -- with ongoing consultation and support check-ins from study clinical staff.
  Interventions: Behavioral: Youth-Nominated Support Team
- Enhanced Treatment as Usual (No Intervention): Adolescents in this condition receive study assessments and risk management services (at time of assessments) only

INTERVENTIONS:
Behavioral: Youth-Nominated Support Team
  Arms: Youth-Nominated Support Team

SUMMARY:
This study will attempt to improve treatment adherence and reduce suicide risk among adolescents who are at risk for attempting suicide.

DETAILED DESCRIPTION:
Despite substantial knowledge about adolescent suicide risk factors, few studies have been conducted to identify effective interventions for suicidal adolescents.

Youth-Nominated Support Team (YST) is an intervention designed to help suicidal adolescents after hospitalization. It is a psychoeducational social network intervention that targets poor treatment adherence and difficulties with social support. YST is designed to be a supplement to traditional or usual treatments.

Participants are randomly assigned to receive either treatment as usual (TAU) or TAU plus YST for 3 months. Adolescents who receive TAU plus YST nominate three or four adults from their family, school, and community settings to function as support persons. The support persons participate in a psychoeducation session that focuses on the adolescent's psychiatric disorder(s), individualized treatment plan, importance of treatment adherence, and suicide risk factors. They also maintain regular contact with the adolescent to support treatment adherence and progress toward treatment goals. Adolescents have assessments at 6 weeks, 3 months, 6 months, and 12 months. Internalizing behavior problems, perceived social support, treatment adherence, adaptive functioning, severity of depression and anxiety, severity and frequency of suicidal thoughts, and suicide attempts are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in a participating psychiatric facility
* Suicidal ideation, intent, or attempt

Exclusion Criteria:

* Severe physical or cognitive impairment that makes informed consent, nominations, or participation in assessments impossible

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 448 (Actual)
Dates: Start 2002-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
suicidal ideation - Suicidal Ideation Questionnaire-JR | 3 month
  Type, frequency, and severity of suicidal thoughts

SECONDARY OUTCOMES:
Depression - Children's Depression Rating Scale-Revised | 3 months

OTHER OUTCOMES:
functional impairment - Child and Adolescent Functional Assessment Scale | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A. King, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- Child and Adolescent Psychiatry Hospital, University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832
- [Derived] King CA, Arango A, Kramer A, Busby D, Czyz E, Foster CE, Gillespie BW; YST Study Team. Association of the Youth-Nominated Support Team Intervention for Suicidal Adolescents With 11- to 14-Year Mortality Outcomes: Secondary Analysis of a Randomized Clinical Trial. JAMA Psychiatry. 2019 May 1;76(5):492-498. doi: 10.1001/jamapsychiatry.2018.4358. PMID 30725077